CLINICAL TRIAL: NCT03094663
Title: Analgesia After Total Knee Arthroplasty: Adductor Canal Block With Periarticular Injection and IPACK (ACB/PAI/IPACK) Versus Periarticular Injection (PAI). A Double-Blinded Randomized Controlled Trial
Brief Title: Adductor Canal Block With Periarticular Injection and IPACK (ACB/PAI/IPACK) Versus Periarticular Injection (PAI)
Acronym: IPACK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-0168
Record Dates: First submitted 2017-02-21; First posted 2017-03-29 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Knee Arthropathy
Keywords: IPACK; PAI
MeSH Terms: interventions — Bupivacaine; Epinephrine; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Cefazolin; Cephalosporins; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peri-Articular Injections only (Active Comparator): Combined spinal epidural anesthetic with 1.5% Mepivacaine (60mg)
  1. Injection prior to cementation
     1. bupivacaine 0.5% with epinephrine 30cc;
     2. methylprednisolone, 40 mg/ml, 1 ml
     3. cefazolin, 500 mg in 10 ml
     4. normal saline, 22cc
  2. Superficial injection prior to closure.
     1. 20cc 0.25% bupivacaine
     2. 2 mg IV dexamethasone.
  Interventions: Drug: Bupivacaine with epinephrine; Drug: Methylprednisolone; Drug: Cefazolin; Device: 8 MHz. Chiba needle; Drug: Bupivacaine 25cc; Drug: Bupivacaine 20cc; Drug: Dexamethasone
- Peri-Articular Injections, Adductor Canal Block, and IPACK (Experimental): Combined spinal epidural anesthetic with 1.5% Mepivacaine (60mg)
  1. Injection prior to cementation
     1. bupivacaine 0.25% with epinephrine 30cc;
     2. methylprednisolone, 40 mg/ml, 1 ml
     3. cefazolin, 500 mg in 10 ml
     4. normal saline, 22cc
  2. Superficial injection prior to closure.
     a. 20cc 0.25% bupivacaine
  3. Adductor canal block technique (supine position, post IV sedation)
     a. Mid-thigh injection of 15 cc of bupivacaine 0.25% with 2 mg of PF Dexamethasone
  4. IPACK technique (supine position) a. 25 cc 0.25% bupivacaine
  Interventions: Drug: Bupivacaine with epinephrine; Drug: Methylprednisolone; Drug: Cefazolin; Device: 8 MHz. Chiba needle; Drug: Bupivacaine with Dexamethasone; Drug: Bupivacaine 25cc; Drug: Bupivacaine 20cc

INTERVENTIONS:
Drug: Bupivacaine with epinephrine — bupivacaine 0.5% with epinephrine 30cc
  Other Names: Sensorcaine/Epinephrine, Sensorcaine-MPF/Epinephrine, Marcaine-Epinephrine (PF)
Drug: Methylprednisolone — 40 mg/ml, 1 ml
  Other Names: Depo-Medrol, Solu-Medrol, Medrol
Drug: Cefazolin — 500 mg in 10 ml
  Other Names: cephalosporin antibiotics
Device: 8 MHz. Chiba needle — 22G/ 4 inches
Drug: Bupivacaine with Dexamethasone — 15 cc of bupivacaine 0.25% with 2 mg of PF Dexamethasone
  Other Names: dexamethasone to non-liposomal bupivacaine
  Arms: Peri-Articular Injections, Adductor Canal Block, and IPACK
Drug: Bupivacaine 25cc — 25 cc 0.25% bupivacaine
  Other Names: Exparel, Marcaine, Marcaine Spinal (PF)
Drug: Bupivacaine 20cc — 20cc 0.25% bupivacaine
  Other Names: Exparel, Marcaine, Marcaine Spinal (PF)
Drug: Dexamethasone — 2 mg IV dexamethasone.
  Other Names: Ozurdex, Maxidex, DexPak 6 Day
  Arms: Peri-Articular Injections only

SUMMARY:
A comparison of two pain control methods - the combination of Adductor Canal Block (ACB)/Periarticular Injection (PAI)/Infiltration of the interspace between the popliteal artery and the capsule of the posterior knee (IPACK) versus the Periarticular Injection (PAI) - in patients undergoing total knee arthroplasty. Primary outcome is NRS pain scores with ambulation on postoperative day one (24 hours post-block administration).

DETAILED DESCRIPTION:
Total knee arthroplasties (TKA) are severely painful surgeries that require optimal pain control to ensure expeditious recovery and discharge. Nerve blocks, such as the femoral and sciatic nerves, are instrumental in effectively providing pain relief and improving patient satisfaction. However, though pain scores notably decreased with the introduction of nerve blocks, motor blockade rendered these patients immobile and may pose a fall risk early in the post-operative period. The advent of ultrasound introduces newer block techniques with adequate analgesia without the cost of motor blockade.

The adductor canal block serves as an alternative to the femoral or sciatic nerve blocks in providing anterior knee analgesia without significantly compromising quadriceps strength. However, patients' posterior knee compartment remains an issue for pain control. Sciatic and posterior tibial nerve blocks were implemented but again, results in motor blockade. A small percentage of sciatic nerve block cases also exhibit foot drop due to peroneal nerve injury. Alternatively, as a sensory block, the periarticular injection (PAI) proves to hasten ambulation and recovery after TKA. The PAI blind injection into the posterior capsule seems to aid in pain control of the posterior compartment and reduces the total number physical therapy sessions.

Injection in the interspace between the Popliteal Artery and Capsule of the posterior Knee (IPACK) provides an alternative to the PAI blind technique for analgesia in the posterior compartment. The IPACK block is not a nerve block, but rather infiltrates the area between the popliteal artery and femur. This area is rich with sensory nerve fibers from the posterior capsule of the knee, which originates from the sciatic and posterior tibial nerve. In this prospective study, we will compare pain scores between the three groups: ACB/PAI/IPACK, ACB/IPACK and PAI only. We will determine whether there is a difference between groups in NRS pain score with ambulation 24 hours post block administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for a primary either partial or total knee arthroplasty with a participating surgeon
* Age 18 to 80 years
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (secondary outcomes include questionnaires validated in English only)
* Patients of participating surgeons

Exclusion Criteria:

* Hepatic or renal insufficiency
* Younger than 18 years old and older than 80
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI > 40
* Diabetes
* ASA of IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months, or daily oral morphine equivalent of >5mg/day for one month)
* Patients with severe valgus deformity and flexion contracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital For Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DH, Beathe JC, Lin Y, YaDeau JT, Maalouf DB, Goytizolo E, Garnett C, Ranawat AS, Su EP, Mayman DJ, Memtsoudis SG. Addition of Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee and Adductor Canal Block to Periarticular Injection Enhances Postoperative Pain Control in Total Knee Arthroplasty: A Randomized Controlled Trial. Anesth Analg. 2019 Aug;129(2):526-535. doi: 10.1213/ANE.0000000000003794. PMID 30234517

RESULTS

PARTICIPANT FLOW:
Groups:
- Peri-Articular Injections Only: Combined spinal epidural anesthetic with 1.5% Mepivacaine (60mg)
  1. Injection prior to cementation
     1. bupivacaine 0.5% with epinephrine 30cc;
     2. methylprednisolone, 40 mg/ml, 1 ml
     3. cefazolin, 500 mg in 10 ml
     4. normal saline, 22cc
  2. Superficial injection prior to closure.
     1. 20cc 0.25% bupivacaine
     2. 2 mg IV dexamethasone.
        Bupivacaine: 0.5% with epinephrine 30cc
        Methylprednisolone: 40 mg/ml, 1 ml
        Cefazolin: 500 mg in 10 ml
        8 MHz. Chiba needle: 22G/ 4 inches
        25 cc 0.25% bupivacaine: 25 cc 0.25% bupivacaine
        20cc 0.25% bupivacaine: 20cc 0.25% bupivacaine
        2 mg IV dexamethasone.: 2 mg IV dexamethasone.
        bupivacaine 0.5% with epinephrine 30cc: bupivacaine 0.5% with epinephrine 30cc
- Peri-Articular Injections, Adductor Canal Block, and IPACK: Combined spinal epidural anesthetic with 1.5% Mepivacaine (60mg)
  1. Injection prior to cementation a. bupivacaine 0.25% with epinephrine 30cc; b. methylprednisolone, 40 mg/ml, 1 ml c. cefazolin, 500 mg in 10 ml d. normal saline, 22cc
  2. Superficial injection prior to closure.
     a. 20cc 0.25% bupivacaine
  3. Adductor canal block technique (supine position, post IV sedation) a. Mid-thigh injection of 15 cc of bupivacaine 0.25% with 2 mg of PF Dexamethasone
  4. IPACK technique (supine position)
     1. 25 cc 0.25% bupivacaine
        Bupivacaine: 0.5% with epinephrine 30cc
        Methylprednisolone: 40 mg/ml, 1 ml
        Cefazolin: 500 mg in 10 ml
        8 MHz. Chiba needle: 22G/ 4 inches
        15 cc of bupivacaine 0.25% with 2 mg of preservative free Dexamethasone: 15 cc of bupivacaine 0.25% with 2 mg of PF Dexamethasone
        25 cc 0.25% bupivacaine: 25 cc 0.25% bupivacaine
        20cc 0.25% bupivacaine: 20cc 0.25% bupivacaine
Period: Overall Study
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Started | 43 | 43
Completed | 43 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.1) | 68.3 (7) | 67.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 13 | 20 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 42 | 39 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 40 | 39 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 86
Height [Mean (Standard Deviation); unit: cm] | 167.6 (10.5) | 168.2 (9.5) | 167.9 (9.9)
Weight [Mean (Standard Deviation); unit: kg] | 84.3 (17.1) | 80.4 (15.9) | 82.4 (16.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (4.8) | 28.3 (4.1) | 29.1 (4.5)
ASA status [Count of Participants; unit: Participants] — The purpose of an ASA score is to assess and communicate a patient's pre-anesthesia medical co-morbidities. Assigning an ASA level is a clinical decision based on multiple factors. While the ASA classification may initially be determined at various times during the preoperative assessment of the patient, the final assignment of ASA is made on the day of anesthesia care by the anesthesiologist after evaluating the patient.
  ASA I: A normal healthy patient. ASA II: A patient with mild systemic disease. ASA III: A patient with severe systemic disease.
  Participants
    ASA I | 1 | 0 | 1
    ASA II | 41 | 40 | 81
    ASA III | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain Scores
Description: Numeric Rating Scale (NRS) Pain scores with ambulation 24 hours post block administration.
  Min = 0, no pain Max = 10, worst imaginable pain
Time Frame: 24 hours post block administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
score on a scale | 5.0 (1.7) | 1.7 (1.4)

2. Secondary Outcome: Opioid Consumption
Description: Opioid consumption at different intervals. Although collected at different time points, the average amount of opioid across all the time points was calculated and reported.
Time Frame: 24 hours on Post-Operative Day 1, 48 hours on Post-Operative Day 2, and 72 hours on Post-Operative Day 3
Measure: Mean (Standard Deviation); unit: oral morphine equivalents (mg)
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
oral morphine equivalents (mg) | 69.1 (79.9) | 40.6 (32.1)

3. Secondary Outcome: Numeric Rating Scale (NRS) Pain Scores at Rest and With Movement
Description: Numeric Rating Scale (NRS) Pain scores at rest and with movement at different intervals Min = 0, no pain Max = 10, worst imaginable pain
  Despite being collected at various times, the average pain score across all time points was calculated and reported.
Time Frame: 24 hours on Post-Operative Day 1, 48 hours on Post-Operative Day 2, and 72 hours on Post-Operative Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
score on a scale | 3.4 (2.1) | 1.2 (1.6)

4. Secondary Outcome: Ambulation Distance During Physical Therapy
Description: The distance patients were able to walked during physical therapy ambulation. Measured in feet.
  The average distance that patients walked at each time point was calculated and reported for the number of participants analyzed.
Time Frame: It will be assessed on 24 hours on Post-Operative Day 1, 48 hours on Post-Operative Day 2, and 72 hours on Post-Operative Day 3
Population: some patients were discharged or unable to ambulate during time point.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
feet
  Post-operative day 0, <24 hours: number analyzed (Participants) | 43 | 42
  Post-operative day 0, <24 hours | 23.2 (26.1) | 25.7 (28.8)
  Post-operative day 1, 24 hours: number analyzed (Participants) | 42 | 43
  Post-operative day 1, 24 hours | 81.1 (61) | 87.7 (46.2)
  Post-operative day 2, 48 hours: number analyzed (Participants) | 32 | 34
  Post-operative day 2, 48 hours | 112 (38.7) | 116.7 (51.7)
  Post-operative day 3, 72 hours: number analyzed (Participants) | 31 | 29
  Post-operative day 3, 72 hours | 106.5 (51.8) | 119.5 (59.9)

5. Secondary Outcome: Level of Patient Satisfaction With Postoperative Pain Management
Description: Patient satisfaction with their postoperative pain management. Measured on a scale of 0 to 10, with 0 meaning extremely dissatisfied and 10 meaning extremely satisfied.
Time Frame: Post-Operative Day 2
Population: Because patients were not reachable for follow-up on post-operative day 2, the total number of participants analyzed for this outcome was reduced.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 36 | 33
score on a scale | 8.8 (1.3) | 9.5 (1.1)

6. Secondary Outcome: Pain Outcomes
Description: The Pain Outcomes (PainOUT) questionnaire was used to assess postoperative pain, psychological variables associated with pain, opioid consumption, satisfaction, and side effects. Scored on 3 scales of 0 to 10, depending on each individual question:
  0 = no pain, 10 = worst pain imaginable 0 = did not interfere, 10 = completely interfered 0 = not at all, 10 = extremely
  Although measured across different timepoints, the average score of all participants was calculated and reported.
Time Frame: Post-Operative Day 1 and Post-Operative Day 2, average across the two time points reported
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 36 | 33
score on a scale | 6.9 (2.1) | 5.6 (2.5)

7. Secondary Outcome: Hospital Length of Stay
Description: The patients' Length of Stay (LOS) at the hospital will be calculate with the time the patient entered the post-operative care unit being the "begin time" and the time patient was discharged being the "end time." The "end time" will differ for each patient depending on which day (post-operative day 1, post-operative day 2, or post-operative day 3) they were discharged.
  The average length of stay for all patients (reported in minutes) will be reported.
Time Frame: Assessed at either: 24 hours on Post-Operative Day 1, 48 hours on Post-Operative Day 2, or 72 hours on Post-Operative Day 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
minutes | 2991 [2874 to 4289] | 3081 [2833 to 4182]

8. Secondary Outcome: Opioid Related Symptom Distress Scale (ORSDS)
Description: ORSDS scores. A lower score is a better outcome. range is 0 to 4.
Time Frame: Post-Operative Day 1 and Post-Operative Day 2
Population: some patients did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
score on a scale
  Post-operative day 1, 24 hrs | 0.4 (0.3) | 0.3 (0.3)
  Post-operative day 2, 48 hrs: number analyzed (Participants) | 36 | 43
  Post-operative day 2, 48 hrs | 0.5 (0.4) | 0.4 (0.4)

9. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr)
Description: This is a patient-reported joint-specific score used to assess outcomes following total knee arthroplasty. Scores range from 0 to 100, with 0 representing total knee disability and 100 representing perfect knee health. Higher score means better outcome.
  The average score for each time point is reported for each arm.
Time Frame: Measured at pre-operation (day of surgery) and 6 weeks post-operation
Population: Because patients were not reachable for follow-up at 6 weeks post-surgery, the total number of participants analyzed for this outcome was reduced.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
Number analyzed (Participants) | 43 | 43
score on a scale
  Pre-operation | 54 (9) | 52 (10)
  6 weeks post surgery: number analyzed (Participants) | 41 | 42
  6 weeks post surgery | 73 (11) | 77 (13)

ADVERSE EVENTS:
Time Frame: Patients were monitored while at the hospital (up to post-operative day 3) and contacted followed up (up to 6-weeks) after their surgery day. Any adverse events that occurred over this time period were documented.
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections, Adductor Canal Block, and IPACK
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03094663/Prot_SAP_000.pdf